CLINICAL TRIAL: NCT00386217
Title: Psychosocial Impact of Cancer-Related Female Infertility
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2003-0568
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Hodgkin's Disease; Cervical Cancer; Breast Cancer; Lymphoma
Keywords: Cervical Cancer; Breast Cancer; Hodgkin's Disease; Non-Hodgkin's Lymphoma; Female Infertility; Telephone Survey
MeSH Terms: conditions — Hodgkin Disease; Uterine Cervical Neoplasms; Breast Neoplasms; Lymphoma; Lymphoma, Non-Hodgkin; Infertility, Female | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Telephone Survey: 90 minute Telephone survey of female cancer survivors
  Interventions: Behavioral: Telephone Survey

INTERVENTIONS:
Behavioral: Telephone Survey — Telephone interview, about 90 minutes, covering demographic information, medical information, health-related quality of life, emotional distress, and stress related to interrupted childbearing.
  Other Names: Questionnaire

SUMMARY:
The success of cancer treatment combined with the trend to delay childbearing is increasing the numbers of women survivors whose childbearing has been interrupted by cancer. For some, treatment has resulted in infertility. Others have been advised to delay pregnancy until a certain follow-up interval or have new fears that pregnancy could be a risk to maternal health. Not least is the concern that children born after a mother's cancer would face increased risks for birth defects or cancer.

The specific aims of this project are as follows:

1. To measure the impact of cancer-related interruption of childbearing on women's long-term emotional well-being and health-related quality of life, over and above other demographic and cancer-related factors
2. To find out if becoming a biological or social mother after cancer treatment decreases the long-term psychosocial impact of interrupted childbearing compared to remaining childless
3. To refine the psychometric properties of questionnaires for female cancer survivors measuring Distress about Cancer-Related Childbearing Issues and Attitudes towards Parenthood after Cancer
4. To define targets for a future intervention to improve female survivors' knowledge about childbearing after cancer, decrease distress associated with interrupted childbearing, and promote peer support.

DETAILED DESCRIPTION:
Women from the M. D. Anderson tumor registry who were diagnosed from 1992 to 1997 with invasive cervical cancer, breast cancer, Hodgkin's disease, or non-Hodgkin's lymphoma will be asked to participate. Researchers have chosen these types of cancers because they are the most common cancers in women of reproductive age. In addition, many of the standard treatments for these diseases have the potential to cause infertility.

If you agree to participate, you will be asked to complete a survey over the phone. Topics that will be addressed by the survey include demographic information (such as age, sex, etc.), medical information, health-related quality of life, emotional distress, and stress related to interrupted childbearing. Some other topics include anxiety related to the impact of cancer on childbearing, menopausal symptoms, spiritual well-being, relationship happiness, sexual satisfaction, and attitudes about parenthood after cancer. The phone survey should take around 90 minutes to complete.

If you feel distressed at any time during or after your participation in this study, you will be given a referral for professional counseling.

THIS IS AN INVESTIGATIONAL STUDY.

Up to 2091 women will be invited to participate in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Women must be survivors of breast cancer, cervical cancer, Hodgkin's Disease, or non-Hodgkin's lymphoma. (We have chosen these three sites because they are the most common malignancies in women of reproductive age that have reasonable rates of long-term survival. In addition, many of the standard treatments for these malignancies impair fertility.)
2. Women must have been diagnosed before the age of 41, i.e., of childbearing age at the time of diagnosis and/or beyond.
3. Women must be at least age 14 currently to participate, because of the concern that younger girls may not be emotionally mature enough to have considered the emotional aspects of infertility, and may also not have full knowledge about reproduction.
4. Women must must have been diagnosed between the years of 1993-1998, making them, roughly 5- to 10-year survivors.
5. We are not going to exclude women based on cancer stage or treatment status, as long as they have survived for 5 to 10 years.

Exclusion Criteria:

1. Women's fluency in English must be adequate to complete the interview (approximately 6th grade level).

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female survivors of breast cancer, cervical cancer, Hodgkin's Disease, or non-Hodgkin's lymphoma, age 14 years and older, who were diagnosed before the age of 41 during the period of 1993-1998.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2004-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Emotional Impact of Cancer Treatment on Childbearing: Female Cancer Survivor Response to Telephone Survey | Single telphone survey lasting about 90 minutes, 4 Years to collect complete surveys

CONTACTS AND LOCATIONS:
Overall Officials: Leslie R. Schover, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org